CLINICAL TRIAL: NCT06980103
Title: Use of a Decision Aid to Resolve Uncertainty About Radioactive Iodine Treatment in Patients With Intermediate Risk Thyroid Cancer: The Radiance Trial
Brief Title: Use of a Decision Aid to Resolve Uncertainty About Radioactive Iodine Treatment in Patients With Intermediate Risk Thyroid Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 7775339; 4UH3DE031248-03 (NIH)
Record Dates: First submitted 2025-04-08; First posted 2025-05-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Cancer
Keywords: Decision Aid; Radioactive Iodine Treatment; Thyroid Cancer; Intermediate Risk; Differentiated Thyroid Cancer; Intermediate risk DTC
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Decision Support Techniques; Iodine-131; Therapeutics

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Condition (Active Comparator): Patients randomized in the Usual Care Condition arm will receive a link for the American Cancer Society website on Radioactive Iodine (Radioiodine) Therapy for Thyroid Cancer as our comparison.
  Interventions: Behavioral: Usual Care
- Decision Aid (Experimental): Patients randomized in the RAI Decision website arm will receive information about intermediate risk DTC; treatment options for intermediate risk DTC following thyroidectomy; clarification of the decision to be made (to have RAI therapy or not); risks and benefits of each treatment option, including potential side effects related to salivary gland damage, lacrimal and nasal symptoms, delay in childbearing; clarification of values and preferences around treatment options; structured guidance around communication with the healthcare team and information to support decision-making about RAI.
  Interventions: Behavioral: Decision Aid

INTERVENTIONS:
Behavioral: Decision Aid — The study intervention is a web-based decision aid (DA) developed by the study team. The Radioactive Iodine Decisions decision aid is designed as an educational tool to help patients have information about Radioactive Iodine and encourage them to talk with their medical team about this treatment decision.
  Arms: Decision Aid
Behavioral: Usual Care — Patients randomized in the Usual Care Condition arm will receive a link for the American Cancer Society website on Radioactive Iodine (Radioiodine) Therapy for Thyroid Cancer as our comparison.
  Other Names: American Cancer Society website on Radioactive Iodine (Radioiodine) Therapy
  Arms: Usual Care Condition

SUMMARY:
The goal of this study is to learn if a decision aid (DA) website helps people with thyroid cancer make informed decisions about radioactive iodine (RAI) treatment. The main questions it aims to answer are: - Does the decision aid help participants understand the risks and benefits of RAI treatment? - Does it help participants make choices that reflect what matters most to them? - How does the decision aid compare to usual care in supporting patients through this decision? Participants who have been recently diagnosed with intermediate-risk differentiated thyroid cancer (DTC) will be randomly assigned to one of two groups. One group will receive a special decision aid website. This site includes detailed information about RAI, short videos, drop-down menus with extra details, exercises to help clarify values, and tools to help patients prepare questions for their doctor. The other group will receive the American Cancer Society (ACS) website. This site gives basic information about RAI but does not include interactive tools and is not specific to intermediate-risk thyroid cancer. Follow up surveys will be sent to the participants periodically, first at the start of the study, and again at 1 week, 4 weeks, and 6 months later.

Researchers will compare how the two groups differ in making informed decisions. The decision aid is meant to support, not replace, a conversation with the medical team. Doctor recommendations remain an important part of treatment decisions.

DETAILED DESCRIPTION:
Background Information Differentiated thyroid cancer (DTC) presents with a spectrum of disease severity, which is associated with varying recurrence rates. Radioactive iodine (RAI) treatment is often considered for moderate to high recurrence risk cases. Patients with low-risk DTC typically have very low recurrence rates, and RAI is generally not used. In contrast, patients with high-risk DTC commonly receive RAI due to a substantial risk of recurrence. The intermediate-risk group experiences uncertainty regarding the potential benefit of RAI in reducing recurrence risk. This study is designed to evaluate the effect of a decision aid (DA) on the decision-making process among patients with intermediate-risk DTC.

Rationale In 2020, an estimated 860,000 individuals in the United States were living as thyroid cancer survivors, with approximately 55% classified as having low-risk disease. Use of RAI in patients with high-risk DTC has been associated with extended survival and reduced recurrence. Among patients with intermediate-risk DTC, 15-year survival rates remain high at 85% to 93%. However, the benefits of RAI in this population may apply only to certain subgroups, such as older individuals or those with larger tumors.

The study intervention consists of a web-based decision aid called RAI Decisions. Eligible patients are randomized to either the DA arm or a usual care (UC) arm. The UC arm receives standard educational material from the American Cancer Society (ACS) website.

Decisions regarding RAI in intermediate-risk DTC are more complex due to several factors: variability in disease severity, limited data on risk and benefit, and differences among physicians and institutions in treatment recommendations and communication practices. Additional factors influencing decision-making may include age, comorbidities, and fertility considerations. Current clinical practice guidelines recommend consideration of RAI in this group, rendering the decision one of personal preference. These guidelines have contributed to a shift away from over treatment of DTC.

RAI usage within the intermediate-risk category is often influenced by disease severity markers (e.g., number of lymph nodes involved, thyroglobulin levels), physician specialty and perceptions, geographic proximity to care, and institutional practices such as multidisciplinary tumor board discussions. Standard of care currently ranges from minimal patient engagement to robust shared decision-making. The decision aid used in this study does not intend to direct or alter clinical decisions regarding RAI use. Instead, it is designed to support informed, value-based decisions through balanced educational content. The decision aid clearly states that it does not provide medical advice and that treatment decisions should be made in consultation with the patient's clinical team.

This research addresses a documented gap in informational support for patients with intermediate-risk DTC making decisions about RAI. The web-based DA seeks to promote informed choice through evidence-based content, interactive tools, and guidance for communicating with healthcare providers. Previous research suggests that patients who understand the trade-offs of treatment options are more likely to make decisions consistent with their values and experience less regret.

Study Design This is a multi-site randomized controlled trial (RCT) conducted at three hospital systems in the Washington, DC metropolitan area. A total of 713 newly diagnosed intermediate-risk DTC patients will be screened to enroll and randomize 408 participants, specifically 204 in the DA arm and 204 in the UC arm. Participants will be assessed at four timepoints: baseline, 1 week, 4 weeks, and 6 months post-randomization. Retention of 85%, calculated as 346 participants, at 6 months is expected.

The primary outcome is informed choice, assessed at 4 weeks. Secondary outcomes include knowledge, decisional conflict, regret, and treatment satisfaction, assessed at 4 weeks and 6 months. Additional analyses will examine whether self-efficacy and satisfaction with physician communication mediate the DA's effect. Exploratory outcomes include quality of life (QOL), treatment choice, and intermediate indicators of cancer recurrence (e.g., serum thyroglobulin levels, lymph node characteristics via ultrasound, and clinician concerns noted during routine care).

Although treatment decisions will be recorded, the DA is not designed to encourage or discourage RAI use. Instead, the focus is on whether patients make informed decisions aligned with their personal values. Because intermediate-risk DTC is generally an indolent condition, the trial will assess surrogate markers of recurrence risk rather than long-term clinical outcomes.

Participants will complete study assessments via phone or online, according to their preference. Assessors will be blinded to randomization status. Satisfaction with the assigned website (DA or UC) will be measured at the end of each follow-up survey. It is hypothesized that the DA will increase rates of informed choice compared to UC among patients with intermediate-risk DTC.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and older
* Patients diagnosed with intermediate risk DTC < 6 months ago and who are making a decision about RAI treatment
* Ability to understand the information conveyed in the informed consent form, pose questions and process answers (e.g., no cognitive impairment per direct consultation with the patient's physician), and, finally, provided informed consent to participate.
* Participants willingness to be contacted and remain available to complete study activities throughout the duration of the study.

Exclusion Criteria:

* Diagnosis of low risk or high risk DTC
* Prior history of RAI
* Clinical contraindications that prevent consideration of RAI (e.g., pregnancy, lactation, neutropenia if considering high dose of RAI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Informed choice about RAI treatment | 4 weeks
  The primary outcome is informed choice measured with the Multi-Dimensional Measure of Informed Choice (MMIC). The scores for informed choice include two components: knowledge categorized as high/low based on the mid-point in the range of scores on the knowledge measure (minimum score of 0 and maximum score of 10; higher scores indicate greater knowledge) and values (attitudes) that are categorized as positive or negative based on the mid-point on the attitude items (minimum score of 4; maximum score of 28; higher scores more greater alignment of the RAI treatment decision with personal values. Informed choice is characterized as informed or uninformed. An informed choice means a decision based on high knowledge and values (attitudes) that align with the patient's preferences and final treatment decision. An uninformed choice occurs when a patient has low knowledge or makes a decision that doesn't match their personal values and attitudes.

SECONDARY OUTCOMES:
Knowledge about RAI | Baseline
  Knowledge about RAI is measured with an adapted version of a knowledge measure developed by Sawka and colleagues, using 10 items with true, false, or unsure response options. Scores range from a minimum of 0 to a maximum of 10. Knowledge refers to a patient's factual understanding of RAI treatment. Higher scores indicate higher knowledge.
Knowledge about RAI | 1 week
  Knowledge about RAI is measured with an adapted version of a knowledge measure developed by Sawka and colleagues, using 10 items with true, false, or unsure response options. Scores range from a minimum of 0 to a maximum of 10. Knowledge refers to a patient's factual understanding of RAI treatment. Higher scores indicate higher knowledge.
Knowledge about RAI | 4 weeks
  Knowledge about RAI is measured with an adapted version of a knowledge measure developed by Sawka and colleagues, using 10 items with true, false, or unsure response options. Scores range from a minimum of 0 to a maximum of 10. Knowledge refers to a patient's factual understanding of RAI treatment. Higher scores indicate higher knowledge.
Knowledge about RAI | 6 months
  Knowledge about RAI is measured with an adapted version of a knowledge measure developed by Sawka and colleagues, using 10 items with true, false, or unsure response options. Scores range from a minimum of 0 to a maximum of 10. Knowledge refers to a patient's factual understanding of RAI treatment. Higher scores indicate higher knowledge.
Decisional Conflict | Baseline
  Decisional Conflict is measured with the 4-item SURE scale, a short form of the Decisional Conflict Scale developed by O'Connor and colleagues. Response options are Yes or No; the minimum score is 0 and the maximum score is 4. Lower scores indicate higher levels of decisional conflict.
Decisional Conflict | 1 week
  Decisional Conflict is measured with the 4-item SURE scale, a short form of the Decisional Conflict Scale developed by O'Connor and colleagues. Response options are Yes or No; the minimum score is 0 and the maximum score is 4. Lower scores indicate higher levels of decisional conflict.
Decisional Conflict | 4 weeks
  Decisional Conflict is measured with the 4-item SURE scale, a short form of the Decisional Conflict Scale developed by O'Connor and colleagues. Response options are Yes or No; the minimum score is 0 and the maximum score is 4. Lower scores indicate higher levels of decisional conflict.
Decisional Conflict | 6 months
  Decisional Conflict is measured with the 4-item SURE scale, a short form of the Decisional Conflict Scale developed by O'Connor and colleagues. Response options are Yes or No; the minimum score is 0 and the maximum score is 4. Lower scores indicate higher levels of decisional conflict.
Decisional Regret | 4 weeks
  Decisional regret is assessed using the 5-item Decisional Regret Scale developed by Brehaut and colleagues. Responses are made on a 5-point Likert Scale from strongly agree to strongly disagree. Scores range from a minimum of 0 to a maximum of 100. Higher scores indicate higher decisional regret.
Decisional Regret | 6 months
  Decisional regret is assessed using the 5-item Decisional Regret Scale developed by Brehaut and colleagues. Responses are made on a 5-point Likert Scale from strongly agree to strongly disagree. Scores range from a minimum of 0 to a maximum of 100. Higher scores indicate higher decisional regret.
Satisfaction with Decision | 6 months
  Satisfaction with treatment decision about RAI treatment is assessed using the 6-item Satisfaction with Decision Scale by Wills and colleagues. Responses are made on a 5-point Likert scale from strongly disagree to strongly agree. Scores range from a minimum of 6 to a maximum of 30. Higher scores indicate higher satisfaction with treatment decision.
Informed choice about RAI treatment | 6 months
  Informed choice is measured with the Multi-Dimensional Measure of Informed Choice (MMIC). The scores for informed choice include two components: knowledge categorized as high/low based on the mid-point in the range of scores on the knowledge measure (minimum score of 0 and maximum score of 10; higher scores indicate greater knowledge) and values (attitudes) that are categorized as positive or negative based on the mid-point on the attitude items (minimum score of 4; maximum score of 28; higher scores more greater alignment of the RAI treatment decision with personal values. Informed choice is characterized as informed or uninformed. An informed choice means a decision based on high knowledge and values (attitudes) that align with the patient's preferences and final treatment decision. An uninformed choice occurs when a patient has low knowledge or makes a decision that doesn't match their personal values and attitudes.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Inova Health System, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No
Upon completion of the study, de-identified data may be shared with other researchers for the purpose of scientific inquiry. We anticipate generating a de-identified dataset to post to a publicly accessible data repository such as Open Science Framework. Prior to posting, requests for access to the de-identified data will be evaluated by the principal investigators and study team to ensure compatibility with the study's objectives and participant confidentiality.

REFERENCES:
- [Background] Mackinnon DP, Lockwood CM, Williams J. Confidence Limits for the Indirect Effect: Distribution of the Product and Resampling Methods. Multivariate Behav Res. 2004 Jan 1;39(1):99. doi: 10.1207/s15327906mbr3901_4. PMID 20157642
- [Background] Kelly KM, Graves KD, Harper FW, Schmidt JE, Dickinson SL, Andrykowski MA. Assessing perceptions of cancer risk: does mode of assessment or numeracy matter? Cancer Detect Prev. 2007;31(6):465-73. doi: 10.1016/j.cdp.2007.10.011. PMID 18061368
- [Background] Ehlers SL, Davis K, Bluethmann SM, Quintiliani LM, Kendall J, Ratwani RM, Diefenbach MA, Graves KD. Screening for psychosocial distress among patients with cancer: implications for clinical practice, healthcare policy, and dissemination to enhance cancer survivorship. Transl Behav Med. 2019 Mar 1;9(2):282-291. doi: 10.1093/tbm/iby123. PMID 30566662
- [Background] Podnos YD, Smith DD, Wagman LD, Ellenhorn JD. Survival in patients with papillary thyroid cancer is not affected by the use of radioactive isotope. J Surg Oncol. 2007 Jul 1;96(1):3-7. doi: 10.1002/jso.20656. PMID 17567872
- [Background] Podnos YD, Smith D, Wagman LD, Ellenhorn JD. Radioactive iodine offers survival improvement in patients with follicular carcinoma of the thyroid. Surgery. 2005 Dec;138(6):1072-6; discussion 1076-7. doi: 10.1016/j.surg.2005.09.021. PMID 16360393
- [Background] Ibrahimpasic T, Nixon IJ, Palmer FL, Whitcher MM, Tuttle RM, Shaha A, Patel SG, Shah JP, Ganly I. Undetectable thyroglobulin after total thyroidectomy in patients with low- and intermediate-risk papillary thyroid cancer--is there a need for radioactive iodine therapy? Surgery. 2012 Dec;152(6):1096-105. doi: 10.1016/j.surg.2012.08.034. PMID 23158181
- [Background] Ghaznavi SA, Ganly I, Shaha AR, English C, Wills J, Tuttle RM. Using the American Thyroid Association Risk-Stratification System to Refine and Individualize the American Joint Committee on Cancer Eighth Edition Disease-Specific Survival Estimates in Differentiated Thyroid Cancer. Thyroid. 2018 Oct;28(10):1293-1300. doi: 10.1089/thy.2018.0186. Epub 2018 Aug 2. PMID 29897011
- [Background] Ruel E, Thomas S, Dinan M, Perkins JM, Roman SA, Sosa JA. Adjuvant radioactive iodine therapy is associated with improved survival for patients with intermediate-risk papillary thyroid cancer. J Clin Endocrinol Metab. 2015 Apr;100(4):1529-36. doi: 10.1210/jc.2014-4332. Epub 2015 Feb 2. PMID 25642591
- [Background] Yang Z, Flores J, Katz S, Nathan CA, Mehta V. Comparison of Survival Outcomes Following Postsurgical Radioactive Iodine Versus External Beam Radiation in Stage IV Differentiated Thyroid Carcinoma. Thyroid. 2017 Jul;27(7):944-952. doi: 10.1089/thy.2016.0650. Epub 2017 May 17. PMID 28446057
- [Background] Chow SM, Law SC, Mendenhall WM, Au SK, Chan PT, Leung TW, Tong CC, Wong IS, Lau WH. Papillary thyroid carcinoma: prognostic factors and the role of radioiodine and external radiotherapy. Int J Radiat Oncol Biol Phys. 2002 Mar 1;52(3):784-95. doi: 10.1016/s0360-3016(01)02686-4. PMID 11849802
- [Background] Chow SM, Yau S, Kwan CK, Poon PC, Law SC. Local and regional control in patients with papillary thyroid carcinoma: specific indications of external radiotherapy and radioactive iodine according to T and N categories in AJCC 6th edition. Endocr Relat Cancer. 2006 Dec;13(4):1159-72. doi: 10.1677/erc.1.01320. PMID 17158761
- [Background] Jonklaas J, Sarlis NJ, Litofsky D, Ain KB, Bigos ST, Brierley JD, Cooper DS, Haugen BR, Ladenson PW, Magner J, Robbins J, Ross DS, Skarulis M, Maxon HR, Sherman SI. Outcomes of patients with differentiated thyroid carcinoma following initial therapy. Thyroid. 2006 Dec;16(12):1229-42. doi: 10.1089/thy.2006.16.1229. PMID 17199433
- [Background] Grani G, Zatelli MC, Alfo M, Montesano T, Torlontano M, Morelli S, Deandrea M, Antonelli A, Francese C, Ceresini G, Orlandi F, Maniglia CA, Bruno R, Monti S, Santaguida MG, Repaci A, Tallini G, Fugazzola L, Monzani F, Giubbini R, Rossetto R, Mian C, Crescenzi A, Tumino D, Pagano L, Pezzullo L, Lombardi CP, Arvat E, Petrone L, Castagna MG, Spiazzi G, Salvatore D, Meringolo D, Solaroli E, Monari F, Magri F, Triggiani V, Castello R, Piazza C, Rossi R, Ferraro Petrillo U, Filetti S, Durante C. Real-World Performance of the American Thyroid Association Risk Estimates in Predicting 1-Year Differentiated Thyroid Cancer Outcomes: A Prospective Multicenter Study of 2000 Patients. Thyroid. 2021 Feb;31(2):264-271. doi: 10.1089/thy.2020.0272. Epub 2020 Jul 1. PMID 32475305
- [Background] Tuttle RM, Haddad RI, Ball DW, Byrd D, Dickson P, Duh QY, Ehya H, Haymart M, Hoh C, Hunt JP, Iagaru A, Kandeel F, Kopp P, Lamonica DM, Lydiatt WM, McCaffrey J, Moley JF, Parks L, Raeburn CD, Ridge JA, Ringel MD, Scheri RP, Shah JP, Sherman SI, Sturgeon C, Waguespack SG, Wang TN, Wirth LJ, Hoffmann KG, Hughes M. Thyroid carcinoma, version 2.2014. J Natl Compr Canc Netw. 2014 Dec;12(12):1671-80; quiz 1680. doi: 10.6004/jnccn.2014.0169. PMID 25505208
- [Background] Carhill AA, Litofsky DR, Ross DS, Jonklaas J, Cooper DS, Brierley JD, Ladenson PW, Ain KB, Fein HG, Haugen BR, Magner J, Skarulis MC, Steward DL, Xing M, Maxon HR, Sherman SI. Long-Term Outcomes Following Therapy in Differentiated Thyroid Carcinoma: NTCTCS Registry Analysis 1987-2012. J Clin Endocrinol Metab. 2015 Sep;100(9):3270-9. doi: 10.1210/JC.2015-1346. Epub 2015 Jul 14. PMID 26171797
- [Background] Wallner LP, Reyes-Gastelum D, Hamilton AS, Ward KC, Hawley ST, Haymart MR. Patient-Perceived Lack of Choice in Receipt of Radioactive Iodine for Treatment of Differentiated Thyroid Cancer. J Clin Oncol. 2019 Aug 20;37(24):2152-2161. doi: 10.1200/JCO.18.02228. Epub 2019 Jul 8. PMID 31283406
- [Background] Sawka AM, Rilkoff H, Tsang RW, Brierley JD, Rotstein L, Ezzat S, Asa SL, Segal P, Kelly C, Zahedi A, Gafni A, Goldstein DP. The rationale of patients with early-stage papillary thyroid cancer for accepting or rejecting radioactive iodine remnant ablation. Thyroid. 2013 Feb;23(2):246-7. doi: 10.1089/thy.2012.0422. No abstract available. PMID 23009127
- [Background] Sawka AM, Straus S, Gafni A, Meiyappan S, David D, Rodin G, Brierley JD, Tsang RW, Thabane L, Rotstein L, Ezzat S, Goldstein DP. Thyroid cancer patients' involvement in adjuvant radioactive iodine treatment decision-making and decision regret: an exploratory study. Support Care Cancer. 2012 Mar;20(3):641-5. doi: 10.1007/s00520-011-1302-x. Epub 2011 Nov 10. PMID 22072050
- [Background] Sawka AM, Straus S, Rodin G, Tsang RW, Brierley JD, Rotstein L, Segal P, Gafni A, Ezzat S, Goldstein DP. Exploring the relationship between patients' information preference style and knowledge acquisition process in a computerized patient decision aid randomized controlled trial. BMC Med Inform Decis Mak. 2015 Jun 19;15:48. doi: 10.1186/s12911-015-0168-0. PMID 26088605
- [Background] Sawka AM, Straus S, Rodin G, Thorpe KE, Ezzat S, Gafni A, Goldstein DP. Decision aid on radioactive iodine treatment for early stage papillary thyroid cancer: update to study protocol with follow-up extension. Trials. 2015 Jul 14;16:302. doi: 10.1186/s13063-015-0819-6. PMID 26169592
- [Background] Shay LA, Lafata JE. Where is the evidence? A systematic review of shared decision making and patient outcomes. Med Decis Making. 2015 Jan;35(1):114-31. doi: 10.1177/0272989X14551638. Epub 2014 Oct 28. PMID 25351843
- [Background] Stacey D, Legare F, Lewis K, Barry MJ, Bennett CL, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2017 Apr 12;4(4):CD001431. doi: 10.1002/14651858.CD001431.pub5. PMID 28402085
- [Background] Barry MJ, Edgman-Levitan S. Shared decision making--pinnacle of patient-centered care. N Engl J Med. 2012 Mar 1;366(9):780-1. doi: 10.1056/NEJMp1109283. No abstract available. PMID 22375967
- [Background] Scholl I, Hahlweg P, Lindig A, Bokemeyer C, Coym A, Hanken H, Muller V, Smeets R, Witzel I, Kriston L, Harter M. Evaluation of a program for routine implementation of shared decision-making in cancer care: study protocol of a stepped wedge cluster randomized trial. Implement Sci. 2018 Mar 27;13(1):51. doi: 10.1186/s13012-018-0740-y. PMID 29580249
- [Background] Elwyn G, Frosch DL, Kobrin S. Implementing shared decision-making: consider all the consequences. Implement Sci. 2016 Aug 8;11:114. doi: 10.1186/s13012-016-0480-9. PMID 27502770
- [Background] Beers E, Lee Nilsen M, Johnson JT. The Role of Patients: Shared Decision-Making. Otolaryngol Clin North Am. 2017 Aug;50(4):689-708. doi: 10.1016/j.otc.2017.03.006. Epub 2017 May 30. PMID 28571664
- [Background] Chewning B, Bylund CL, Shah B, Arora NK, Gueguen JA, Makoul G. Patient preferences for shared decisions: a systematic review. Patient Educ Couns. 2012 Jan;86(1):9-18. doi: 10.1016/j.pec.2011.02.004. Epub 2011 Apr 6. PMID 21474265
- [Background] Clayman ML, Bylund CL, Chewning B, Makoul G. The Impact of Patient Participation in Health Decisions Within Medical Encounters: A Systematic Review. Med Decis Making. 2016 May;36(4):427-52. doi: 10.1177/0272989X15613530. Epub 2015 Nov 19. PMID 26585293
- [Background] Moore MD, Postma E, Gray KD, Ullmann TM, Hurley JR, Goldsmith S, Sobel VR, Schulman A, Scognamiglio T, Christos PJ, Hassett E, Luick J, Whitehall D, Zarnegar R, Fahey TJ 3rd. Less is More: The Impact of Multidisciplinary Thyroid Conference on the Treatment of Well-Differentiated Thyroid Carcinoma. World J Surg. 2018 Feb;42(2):343-349. doi: 10.1007/s00268-017-4308-9. PMID 29058064
- [Background] Papaleontiou M, Banerjee M, Yang D, Sisson JC, Koenig RJ, Haymart MR. Factors that influence radioactive iodine use for thyroid cancer. Thyroid. 2013 Feb;23(2):219-24. doi: 10.1089/thy.2012.0380. PMID 23134514
- [Background] Jacobs D, Breen CT, Pucar D, Holt EH, Judson BL, Mehra S. Changes in Population-Level and Institutional-Level Prescribing Habits of Radioiodine Therapy for Papillary Thyroid Cancer. Thyroid. 2021 Feb;31(2):272-279. doi: 10.1089/thy.2020.0237. Epub 2020 Sep 22. PMID 32811347
- [Background] Sacks W, Wong RM, Bresee C, Braunstein GD. Use of evidence-based guidelines reduces radioactive iodine treatment in patients with low-risk differentiated thyroid cancer. Thyroid. 2015 Apr;25(4):377-85. doi: 10.1089/thy.2014.0298. Epub 2015 Feb 6. PMID 25578116
- [Background] Haymart MR, Banerjee M, Yang D, Stewart AK, Sisson JC, Koenig RJ, Doherty GM, Griggs JJ. Variation in the management of thyroid cancer. J Clin Endocrinol Metab. 2013 May;98(5):2001-8. doi: 10.1210/jc.2012-3355. Epub 2013 Mar 28. PMID 23539722
- [Background] Marti JL, Morris LGT, Ho AS. Selective use of radioactive iodine (RAI) in thyroid cancer: No longer "one size fits all". Eur J Surg Oncol. 2018 Mar;44(3):348-356. doi: 10.1016/j.ejso.2017.04.002. Epub 2017 May 3. PMID 28545679
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Jonklaas J, Carr AL, Luta G, Yu C, Jensen RE, Reasner E, Winslow J, Kuo CC, Davidson BJ, Esposito G, Bloom G, Diamond-Rossi SA, Graves KD. Salivary, lacrimal and nasal (SALANS) measure to assess side effects following radioactive iodine treatment: development, psychometric properties, and factor structure. Qual Life Res. 2024 Jul;33(7):2011-2023. doi: 10.1007/s11136-024-03684-2. Epub 2024 May 20. PMID 38769210
- [Background] Melhem SJ, Nabhani-Gebara S, Kayyali R. Digital Trends, Digital Literacy, and E-Health Engagement Predictors of Breast and Colorectal Cancer Survivors: A Population-Based Cross-Sectional Survey. Int J Environ Res Public Health. 2023 Jan 13;20(2):1472. doi: 10.3390/ijerph20021472. PMID 36674237
- [Background] Edelen MO, Zeng C, Hays RD, Rodriguez A, Hanmer J, Baumhauer J, Cella D, Reeve BB, Herman PM. Development of an ultra-short measure of eight domains of health-related quality of life for research and clinical care: the patient-reported outcomes measurement information system(R) PROMIS(R)-16 profile. Qual Life Res. 2025 Jan;34(1):3-15. doi: 10.1007/s11136-023-03597-6. Epub 2024 Feb 6. PMID 38319489
- [Background] Marteau TM, Dormandy E, Michie S. A measure of informed choice. Health Expect. 2001 Jun;4(2):99-108. doi: 10.1046/j.1369-6513.2001.00140.x. PMID 11359540
- [Background] Chew LD, Griffin JM, Partin MR, Noorbaloochi S, Grill JP, Snyder A, Bradley KA, Nugent SM, Baines AD, Vanryn M. Validation of screening questions for limited health literacy in a large VA outpatient population. J Gen Intern Med. 2008 May;23(5):561-6. doi: 10.1007/s11606-008-0520-5. Epub 2008 Mar 12. PMID 18335281
- [Background] Schwartz LM, Woloshin S, Black WC, Welch HG. The role of numeracy in understanding the benefit of screening mammography. Ann Intern Med. 1997 Dec 1;127(11):966-72. doi: 10.7326/0003-4819-127-11-199712010-00003. PMID 9412301
- [Background] Elwyn G, Barr PJ, Grande SW, Thompson R, Walsh T, Ozanne EM. Developing CollaboRATE: a fast and frugal patient-reported measure of shared decision making in clinical encounters. Patient Educ Couns. 2013 Oct;93(1):102-7. doi: 10.1016/j.pec.2013.05.009. Epub 2013 Jun 12. PMID 23768763
- [Background] Arora NK, Weaver KE, Clayman ML, Oakley-Girvan I, Potosky AL. Physicians' decision-making style and psychosocial outcomes among cancer survivors. Patient Educ Couns. 2009 Dec;77(3):404-12. doi: 10.1016/j.pec.2009.10.004. Epub 2009 Nov 4. PMID 19892508
- [Background] Wills CE, Holmes-Rovner M. Preliminary validation of the Satisfaction With Decision scale with depressed primary care patients. Health Expect. 2003 Jun;6(2):149-59. doi: 10.1046/j.1369-6513.2003.00220.x. PMID 12752743
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Sawka AM, Straus S, Rotstein L, Brierley JD, Tsang RW, Asa S, Segal P, Kelly C, Zahedi A, Freeman J, Solomon P, Anderson J, Thorpe KE, Gafni A, Rodin G, Goldstein DP. Randomized controlled trial of a computerized decision aid on adjuvant radioactive iodine treatment for patients with early-stage papillary thyroid cancer. J Clin Oncol. 2012 Aug 10;30(23):2906-11. doi: 10.1200/JCO.2011.41.2734. Epub 2012 Jul 2. PMID 22753906
- [Background] Michie S, Dormandy E, Marteau TM. The multi-dimensional measure of informed choice: a validation study. Patient Educ Couns. 2002 Sep;48(1):87-91. doi: 10.1016/s0738-3991(02)00089-7. PMID 12220754
- See also: American Cancer Society. Radioactive Iodine (radioiodine) Therapy for Thyroid Cancer. — https://www.cancer.org/cancer/thyroid-cancer/treating/radioactive-iodine.html
- See also: NCCN Guidelines. NCCN Guidelines Version 1.2024 Distress Management — https://www.nccn.org/docs/default-source/patient-resources/nccn_distress_thermometer